CLINICAL TRIAL: NCT02735213
Title: A Prospective Non-inferiority Study of the Use of Micropulse 577nm Laser vs Traditional Laser Treatment in Central Serous Chorioretinopathy
Brief Title: Micropulse 577nm Laser vs Traditional Laser Treatment in Central Serous Chorioretinopathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiaoling Liu, professor, The Eye Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-2016005
Record Dates: First submitted 2016-03-16; First posted 2016-04-12 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Central Serous Choroidopathy
Keywords: Central Serous Choroidopathy; Micropulse Laser Treatment; Traditional laser Treatment; optical coherence tomography
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 577-MPL (Experimental): 577nm subthreshold micropulse laser(577-MPL) will be performed on the areas identified on hyperfluorescent "hot spots" on the mid-phase (3 minutes) fluorescein. Multiple laser spots will be applied, covering the leakage area. Retreatment will be given in 12 weeks If SRF is not completely absorbed and CRT>= 250um.
  Interventions: Device: 577-MPL
- TLT (Active Comparator): Traditional laser will be performed of the areas identified on hyperfluorescent "hot spots" on the mid-phase (3 minutes) fluorescein.Traditional laser spots will be applied, covering the leakage area. Retreatment will be given in 12 weeks If SRF is not completely absorbed and CRT>= 250um.
  Interventions: Device: TLT

INTERVENTIONS:
Device: 577-MPL — 9 spots multispot micropulse mode(without spacing between the spots),160 um spot size, 0.2 second duration, 5% duty cycle(ON time 0.1ms + OFF time 1.9ms), and 250~400 milliWatts of power(50% threshold power),150~200 spots, the laser area is the corresponding leakage on mid-phase FA and around leakage.
  Arms: 577-MPL
Device: TLT — contimuous wave,100um spot size, 0.05 seconds duration, 55~60 milliwatts of power, 18~27 spots,the laser area is the corresponding leakage on mid-phase FA.
  Arms: TLT

SUMMARY:
The purpose of this study is to observe whether micropulse laser (MPL) is noninferiority to traditional laser therapy in central serous chorioretinopathy.

DETAILED DESCRIPTION:
Central serous chorioretinopathy (CSC) is characterized by serous detachment of neurosensory retina which can cause lose in visual acuity. Some studies have shown that traditional laser treatment (TLT) is effective on CSC, although accompanied with side-effects, such as scar. Recent retrospective studies suggest micropulse laser (MPL) therapy may also be effective without obvious complications in this disease. But to date, there is no study on effectiveness of CSC between TLT and MPL.

The study is the first prospective randomized controlled trial about 577nm micropulse laser versus traditional laser treatment in central serous chorioretinopathy. It is a noninferiority study. The investigators hypothesize that application of 577nm micropulse laser in patients with CSC will prompt resolution of CSC as measured by ocular coherence tomography and best corrected visual acuity.This will be a pilot study to establish sound methods and provide some insights to the safety and efficacy of CSC treatment. The primary outcome measures is the change of BCVA in 12 week.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CSC；
2. age>=18 years old;
3. Duration is less than 6 months；
4. the presence of subretinal fluid(SRF) involving the macula and detected by use of optical coherence tomography (OCT), and CRT>=250um;
5. active leakage located at ring 2 and ring 3 (ETDRS rings) on fluorescein angiography (FA).

Exclusion Criteria:

1. Patients with no case of CSC；
2. Patients with other macular comorbidities including but not limited to diabetic retinopathy, macular degeneration；
3. Patients with prior retinal treatment less than 3 months；
4. Inability to obtain photographs or to perform FA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change of Best Corrected Visual Acuity (BCVA) | 12 week
  ETDRS BCVA

SECONDARY OUTCOMES:
the number of patients without any subretinal fluid (SRF) | 3 week, 7 week, 12 week
  SRF
Change of the central retinal thickness (CRT) | 3 week, 7 week, 12 week
  CRT
laser scar in area lasered on | 12 week
  colour image and OCT infared image
the number of patients need retreatment | 12 week
  PRN (pro re nata), only for SRF not completely absorbed and CRT >=250um

CONTACTS AND LOCATIONS:
Locations (1):
- The eye of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] Salehi M, Wenick AS, Law HA, Evans JR, Gehlbach P. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2015 Dec 22;2015(12):CD011841. doi: 10.1002/14651858.CD011841.pub2. PMID 26691378
- [Background] Iacono P, Battaglia Parodi M, Falcomata B, Bandello F. Central Serous Chorioretinopathy Treatments: A Mini Review. Ophthalmic Res. 2015;55(2):76-83. doi: 10.1159/000441502. Epub 2015 Dec 1. PMID 26619293
- [Background] Daruich A, Matet A, Dirani A, Bousquet E, Zhao M, Farman N, Jaisser F, Behar-Cohen F. Central serous chorioretinopathy: Recent findings and new physiopathology hypothesis. Prog Retin Eye Res. 2015 Sep;48:82-118. doi: 10.1016/j.preteyeres.2015.05.003. Epub 2015 May 27. PMID 26026923
- [Background] Loo RH, Scott IU, Flynn HW Jr, Gass JD, Murray TG, Lewis ML, Rosenfeld PJ, Smiddy WE. Factors associated with reduced visual acuity during long-term follow-up of patients with idiopathic central serous chorioretinopathy. Retina. 2002 Feb;22(1):19-24. doi: 10.1097/00006982-200202000-00004. PMID 11884873
- [Background] Ficker L, Vafidis G, While A, Leaver P. Long-term follow-up of a prospective trial of argon laser photocoagulation in the treatment of central serous retinopathy. Br J Ophthalmol. 1988 Nov;72(11):829-34. doi: 10.1136/bjo.72.11.829. PMID 3061449